CLINICAL TRIAL: NCT04349774
Title: A Prospective, Randomized, Double-Blind, Active-Comparator, Pilot Study to Observe Relative Efficacy of Ultrasound-Guided Erector Spinae Plane Block (ESP) vs. Combination of Ultrasound - Guided Erector Spinae Plane Block With Serratus Anterior Plane Block in Managing Post-operative Pain Following Thoracic Surgery.
Brief Title: Erector Spinae Plane Block vs Erector Spinae Plane Block With Serratus Anterior Plane Block in Thoracic Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never initiated due to COVID-19
Sponsor: Anna Uskova (Other)
Responsible Party: Sponsor-Investigator, Anna Uskova, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19090184
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pain, Postoperative
Keywords: Erector Spinae Plane block; Serratus Anterior Plane block; Thoracic Surgery; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Continuous Erector Spinae Plane block with 20ml 0.375% Bupivacaine and continuous infusion of 0.25% Lidocaine @ 12ml/hr, with single shot Serratus Anterior Plane block with 20ml 0.375% Bupivacaine
  Interventions: Drug: Control Group - ESP block with SAP block
- Treatment Group (Active Comparator): Continuous Erector Spinae Plane block with 20ml 0.375% Bupivacaine and continuous infusion of 0.25% Lidocaine @ 12ml/hr, with single shot Serratus Anterior Plane block with 20ml Normal Saline.
  Interventions: Drug: Treatment Group - ESP block with SAP normal saline

INTERVENTIONS:
Drug: Control Group - ESP block with SAP block — None - Control Group
  Other Names: ESP block with SAP block
  Arms: Control Group
Drug: Treatment Group - ESP block with SAP normal saline — Substitution of normal saline in place of 0.375% Bupivacaine in SAP block
  Other Names: ESP block with SAP normal saline
  Arms: Treatment Group

SUMMARY:
This pilot study will prospectively compare continuous Erector Spinae Plane block (ESP) versus combination of continuous Erector Spinae Plane block and single shot Serratus Anterior Plane block for post-operative pain management in subjects undergoing primary thoracic surgery.

DETAILED DESCRIPTION:
Once consented, the patient will be randomized by computer generated random number to one of the two treatment groups.

Blinding Plan: At the acute pain management office, one member of the research team will be responsible for providing the anesthesiologist in charge of performing the block with a sealed envelope. Each envelope will be labeled with a number corresponding to a matching number labeled on each patient binder. This envelope will contain the randomized block to be administered - ESP with SAP or ESP with SAP normal saline. Once the anesthesiologist knows which block combination to administer, he/she will reseal the envelope and return it to the research team member. This process allows only the anesthesiologist performing the block to have knowledge of the block being administered, keeping both the patients and research team members blinded. The envelopes and binders will be kept by the principle investigator in a safe place and only reopened to be analyzed at the end of the study.

All study procedures will take place in the preoperative patient room in DAS prior to surgery, as is standard practice in this institution. The consent process will take place prior to performing any research procedures.

If randomized to the ESP block with SAP normal saline, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach: Prior to initiating the block procedure and receiving any sedative medications, patient will be asked to give 3 maximum efforts using the incentive spirometer by first taking a maximum breath in and blowing out forcefully and completely into the incentive spirometer device. Average of these three efforts will be recorded as the patient's incentive spirometer effort baseline. Patient will be positioned in seated position with side to be blocked marked. T5 spinous process will be identified by palpating starting with C7 and continuing caudad. C7 is the most prominent spinous process anatomically. T5 spinous process will be marked with a marking pen. Block area will be cleaned using 2% Chlorhexidine solution. Entire block procedure is performed under strict aseptic technique. Ultrasound probe covered in sterile probe cover will be placed at the T5 spinous process in a cephalad to caudad orientation and moved lateral until the T5 transverse process is identified. 1-2ml of 1% lidocaine will be administered just above the ultrasound probe for local skin infiltration. An 18 gauge Touhy needle will then be inserted in plane in a cephalad to caudad direction under ultrasound visualization until the tip of the needle touches the T5 transverse process. The T5 transverse process is the anatomical target for this block. 20ml of 0.375% bupivacaine will then be injected using slow fractionated injection, aspirating every 5ml to ensure needle tip is not intravascular. Local anesthetic spread in the appropriate plane will be confirmed with ultrasound. Once injection is complete, a 20 gauge non-stimulating catheter will be inserted through the Touhy needle. Catheter tip placement will be confirmed with ultrasound.

SAP Approach with normal saline - Patient will be placed in a lateral position with the side to be blocked facing up. After disinfecting the block area with 2% Chlorhexidine solution and under strict aseptic technique the ultrasound probe will be placed over the midclavicular region of the thorax in a sagittal plane. Ribs will be counted inferiorly and laterally starting with the 2nd rib, until 5th rib is identified in midaxillary line. At this level the 3 appropriate muscle layers overlying the 5th rib are easily identifiable. Latissimus dorsi M. is superficial and posterior, teres major m. is superior, and serratus m. is deep and inferior. Skin at the block site will be infiltrated with 1-2ml of 1% lidocaine, and a 20 gauge Touhy needle will be introduced in plane under ultrasound visualization in a superoanterior to posteroinferior direction just above the Serratus m. At this point 20ml Normal Saline will be injected using slow fractionated injection, aspirating every 5ml to ensure needle tip is not intravascular. Injectate spread in the appropriate plane will be confirmed with ultrasound. Total procedure time for both injections is expected to take 30 minutes from start to finish.

If randomized to the ESP+SAP block, an anesthesiologist on the Acute Interventional Perioperative Pain Service (AIPPS) will administer the block with this approach: Incentive spirometer effort as described above. ESP performed as described above. SAP block: Patient will be placed in a lateral position with the side to be blocked facing up. After disinfecting the block area with 2% Chlorhexidine solution and under strict aseptic technique the ultrasound probe will be placed over the midclavicular region of the thorax in a sagittal plane. Ribs will be counted inferiorly and laterally starting with the 2nd rib, until 5th rib is identified in midaxillary line. At this level the 3 appropriate muscle layers overlying the 5th rib are easily identifiable. Latissimus dorsi M. is superficial and posterior, teres major m. is superior, and serratus m. is deep and inferior. Skin at the block site will be infiltrated with 1-2ml of 1% lidocaine, and a 20 gauge Touhy needle will be introduced in plane under ultrasound visualization in a superio-anterior to posterio-inferior direction just above the Serratus m. At this point 20ml 0.375% Bupivacaine will be injected using slow fractionated injection, aspirating every 5ml to ensure needle tip is not intravascular. Local anesthetic spread in the appropriate plane will be confirmed with ultrasound. Total procedure time for both injections is expected to take 30 minutes from start to finish.

For ESP block and SAP with normal saline, the local anesthetic used will be 20ml 0.375% bupivacaine for ESP block. ESP block group will also receive SAP block with 20ml Normal Saline. For ESP + SAP block group, the local anesthetic used will be 20ml 0.375% Bupivacaine for ESP block. Local anesthetic used for SAP block will be 20ml 0.375% Bupivacaine.

Anesthetic Management: Both treatment groups will receive the standard anesthetic technique and multimodal analgesic technique including preoperative Gabapentin 300mg PO and Acetaminophen 1000mg PO, intraoperative IV propofol infusion-based general anesthetic combined with sub-anesthetic dose IV ketamine infusion, IV dexmedetomidine infusion, IV acetaminophen, and strict avoidance of intraoperative opioids. Post-operative pain management will also follow standard protocol, using IV hydromorphone (0.2 mg) and PO oxycodone (5-10 mg) on request by patient for moderate to severe pain (NRS >5), IV ketamine infusion 5mg/hr for 48 hours, scheduled acetaminophen 1000mg IV for 24hours.

For study participants, the investigator placing the block will record in the narrative that "this patient is a study participant and received Paravertebral block with ESP approach and SAP block". By documenting the blocks in this way, the research team member collecting the data and the nurses documenting the pain scores will be blinded to whether patient received ESP block with 0.375% Bupivacaine + SAP block with normal saline, or ESP block with 0.375% Bupivacaine + SAP block with 0.375% Bupivacaine.

After surgery, the patient will be followed by the blinded research team for incidence of adverse events, as well as the collection of the primary and secondary outcome measures. These include total narcotic medication consumption, reported as total Morphine equivalent in 24 hours after surgery as primary outcome measures. Secondary outcome measures include pain scores at 6, 12, and 24 hours after surgery, total dose of local anesthetic administered at 12 hours and 24 hours after surgery - reported in (mg), percent change from baseline using incentive spirometer at 6 and 24 hours after block performance, total hospital length of stay - from admission to discharge, and incidence of adverse effects - nausea and vomiting requiring treatment, hypotension, and bradycardia or tachycardia. Pain assessment will be done by nurses in the PACU and on the floor using Numeric Pain Rating Scale, with 0 meaning no pain and 10 meaning worst possible pain. Narcotic medication consumption, pain scores, local anesthetic medication consumption, incentive spirometer values, and adverse effects will be recorded on worksheets included in patient research folders, with each study participant having their own research folder identified only by randomly assigned patient study number. Both nursing staff and research staff (study coordinators) collecting data will remain blinded to whether patient received ESP block with 0.375% Bupivacaine + SAP block with normal saline, or ESP block with 0.375% Bupivacaine + AP block with 0.375% Bupivacaine. Only nurses and study coordinators, not acute pain physicians, will record this data.

Patients in both study groups will receive a nerve block, either ESP alone or ESP & SAP. Both ESP and SAP nerve blocks have an identical side effect profile, and adverse events resulting from administration of either of these blocks would be treated in an identical manner. In light of this, we do not anticipate implementing emergency unblinding of patients. However, in the case of adverse event/s occurring, emergency unblinding procedures will be the following. The principle investigator or co-investigators will be contacted and provided the patient unique study ID number, which will be used to access the master list, which includes patient study ID and the type of block received. The patient will be treated for adverse events pertaining to receiving a nerve block and/or other medications mentioned as part of the research protocol. The patient will then be removed from the study, and no further data collection will occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years old
* Primary Unilateral Thoracic Surgery
* BMI 20 - 36, weight > or = to 50kg
* Male and Female
* All races

Exclusion Criteria:

* Patient refusal
* Inpatient status at time of surgery
* ASA class > or = 4
* Bilateral thoracic surgery
* Pregnancy
* Non-English speaking or inability to participate in the study
* Patients with coagulopathy or on therapeutic anticoagulation
* Chronic Steroid Use
* Narcotic Addiction
* Patients with contraindication to performing either block - active infection at block site, systemic infection, allergy to local anesthetic medications
* Patients undergoing second surgery or urgent/emergent surgery
* Patients weighing <50kg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Total narcotic medication consumption 24 hours after surgery | 24 hours after surgery
  Total narcotic medication consumption - reported as total Morphine equivalent 24 hours after surgery

SECONDARY OUTCOMES:
Pain score after surgery | 6,12, and 24 hours after surgery
  Pain scores measured on a 0-10 scale
Total dose of local anesthetic medication administered after surgery | 12 and 24 hours after surgery
  Total dose of local anesthetic medication received following surgery - reported in (mg)
Percent change from baseline using incentive spirometer after nerve block administration | 6,12,and 24 hours after nerve block administration
  Percent change in incentive spirometer value from baseline
Total length of hospital stay | up to one month
  Total length of hospital stay
Incidence of adverse effects | up to one month
  Nausea, vomiting, hypotension, bradycardia, tachycardia requiring treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Gromov, DO, Principal Investigator — University of Pittsburgh Medical Center; Anna Uskova, MD, Study Director — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center (UPMC) Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Background] Baidya DK, Khanna P, Maitra S. Analgesic efficacy and safety of thoracic paravertebral and epidural analgesia for thoracic surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2014 May;18(5):626-35. doi: 10.1093/icvts/ivt551. Epub 2014 Jan 31. PMID 24488821
- [Background] Bang S, Chung K, Chung J, Yoo S, Baek S, Lee SM. The erector spinae plane block for effective analgesia after lung lobectomy: Three cases report. Medicine (Baltimore). 2019 Jul;98(29):e16262. doi: 10.1097/MD.0000000000016262. PMID 31335674
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Chin KJ. Thoracic wall blocks: From paravertebral to retrolaminar to serratus to erector spinae and back again - A review of evidence. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):67-77. doi: 10.1016/j.bpa.2019.02.003. Epub 2019 Apr 5. PMID 31272655
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Chu GM, Jarvis GC. Serratus Anterior Plane Block to Address Postthoracotomy and Chest Tube-Related Pain: A Report on 3 Cases. A A Case Rep. 2017 Jun 15;8(12):322-325. doi: 10.1213/XAA.0000000000000502. PMID 28614112
- [Background] Cook TM, Riley RH. Analgesia following thoracotomy: a survey of Australian practice. Anaesth Intensive Care. 1997 Oct;25(5):520-4. PMID 9352765
- [Background] Davies RG, Myles PS, Graham JM. A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy--a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2006 Apr;96(4):418-26. doi: 10.1093/bja/ael020. Epub 2006 Feb 13. PMID 16476698
- [Background] Fang B, Wang Z, Huang X. Ultrasound-guided preoperative single-dose erector spinae plane block provides comparable analgesia to thoracic paravertebral block following thoracotomy: a single center randomized controlled double-blind study. Ann Transl Med. 2019 Apr;7(8):174. doi: 10.21037/atm.2019.03.53. PMID 31168455
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Gaio-Lima C, Costa CC, Moreira JB, Lemos TS, Trindade HL. Continuous erector spinae plane block for analgesia in pediatric thoracic surgery: A case report. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):287-290. doi: 10.1016/j.redar.2017.11.010. Epub 2018 Jan 19. English, Spanish. PMID 29370900
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Kelava M, Anthony D, Elsharkawy H. Continuous Erector Spinae Block for Postoperative Analgesia After Thoracotomy in a Lung Transplant Recipient. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):e9-e11. doi: 10.1053/j.jvca.2018.04.041. Epub 2018 Apr 26. No abstract available. PMID 29801724
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192
- [Background] Kim DH, Oh YJ, Lee JG, Ha D, Chang YJ, Kwak HJ. Efficacy of Ultrasound-Guided Serratus Plane Block on Postoperative Quality of Recovery and Analgesia After Video-Assisted Thoracic Surgery: A Randomized, Triple-Blind, Placebo-Controlled Study. Anesth Analg. 2018 Apr;126(4):1353-1361. doi: 10.1213/ANE.0000000000002779. PMID 29324496
- [Background] Kotemane NC, Gopinath N, Vaja R. Analgesic techniques following thoracic surgery: a survey of United Kingdom practice. Eur J Anaesthesiol. 2010 Oct;27(10):897-9. doi: 10.1097/EJA.0b013e32833d1259. PMID 20657297
- [Background] Mayes J, Davison E, Panahi P, Patten D, Eljelani F, Womack J, Varma M. An anatomical evaluation of the serratus anterior plane block. Anaesthesia. 2016 Sep;71(9):1064-9. doi: 10.1111/anae.13549. Epub 2016 Jul 20. PMID 27440171
- [Background] Munoz F, Cubillos J, Bonilla AJ, Chin KJ. Erector spinae plane block for postoperative analgesia in pediatric oncological thoracic surgery. Can J Anaesth. 2017 Aug;64(8):880-882. doi: 10.1007/s12630-017-0894-0. Epub 2017 Apr 26. No abstract available. PMID 28447318
- [Background] Nath S, Bhoi D, Mohan VK, Talawar P. USG-guided continuous erector spinae block as a primary mode of perioperative analgesia in open posterolateral thoracotomy: A report of two cases. Saudi J Anaesth. 2018 Jul-Sep;12(3):471-474. doi: 10.4103/sja.SJA_755_17. PMID 30100851
- [Background] Okmen K, Okmen BM. The efficacy of serratus anterior plane block in analgesia for thoracotomy: a retrospective study. J Anesth. 2017 Aug;31(4):579-585. doi: 10.1007/s00540-017-2364-9. Epub 2017 Apr 26. PMID 28447227
- [Background] Park MH, Kim JA, Ahn HJ, Yang MK, Son HJ, Seong BG. A randomised trial of serratus anterior plane block for analgesia after thoracoscopic surgery. Anaesthesia. 2018 Oct;73(10):1260-1264. doi: 10.1111/anae.14424. Epub 2018 Aug 18. PMID 30120832
- [Background] Piccioni F, Segat M, Falini S, Umari M, Putina O, Cavaliere L, Ragazzi R, Massullo D, Taurchini M, Del Naja C, Droghetti A. Enhanced recovery pathways in thoracic surgery from Italian VATS Group: perioperative analgesia protocols. J Thorac Dis. 2018 Mar;10(Suppl 4):S555-S563. doi: 10.21037/jtd.2017.12.86. PMID 29629202
- [Background] Powell ES, Cook D, Pearce AC, Davies P, Bowler GM, Naidu B, Gao F; UKPOS Investigators. A prospective, multicentre, observational cohort study of analgesia and outcome after pneumonectomy. Br J Anaesth. 2011 Mar;106(3):364-70. doi: 10.1093/bja/aeq379. Epub 2011 Feb 2. PMID 21289374
- [Background] Restrepo-Garces CE, Chin KJ, Suarez P, Diaz A. Bilateral Continuous Erector Spinae Plane Block Contributes to Effective Postoperative Analgesia After Major Open Abdominal Surgery: A Case Report. A A Case Rep. 2017 Dec 1;9(11):319-321. doi: 10.1213/XAA.0000000000000605. PMID 28727597
- [Background] Saad FS, El Baradie SY, Abdel Aliem MAW, Ali MM, Kotb TAM. Ultrasound-guided serratus anterior plane block versus thoracic paravertebral block for perioperative analgesia in thoracotomy. Saudi J Anaesth. 2018 Oct-Dec;12(4):565-570. doi: 10.4103/sja.SJA_153_18. PMID 30429738
- [Background] Shanthanna H, Moisuik P, O'Hare T, Srinathan S, Finley C, Paul J, Slinger P. Survey of Postoperative Regional Analgesia for Thoracoscopic Surgeries in Canada. J Cardiothorac Vasc Anesth. 2018 Aug;32(4):1750-1755. doi: 10.1053/j.jvca.2018.01.003. Epub 2018 Jan 5. PMID 29402627
- [Background] Short HL, Kamalanathan K. Has analgesia changed for lung resection surgery? Anaesthesia. 2018 Apr;73(4):412-416. doi: 10.1111/anae.14188. Epub 2018 Jan 12. No abstract available. PMID 29327465
- [Background] Sihoe AD, Au SS, Cheung ML, Chow IK, Chu KM, Law CY, Wan M, Yim AP. Incidence of chest wall paresthesia after video-assisted thoracic surgery for primary spontaneous pneumothorax. Eur J Cardiothorac Surg. 2004 Jun;25(6):1054-8. doi: 10.1016/j.ejcts.2004.02.018. PMID 15145009
- [Background] Singh S, Chowdhary NK. Erector spinae plane block an effective block for post-operative analgesia in modified radical mastectomy. Indian J Anaesth. 2018 Feb;62(2):148-150. doi: 10.4103/ija.IJA_726_17. No abstract available. PMID 29491525
- [Background] Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Regional analgesia for video-assisted thoracic surgery: a systematic review. Eur J Cardiothorac Surg. 2014 Jun;45(6):959-66. doi: 10.1093/ejcts/ezt525. Epub 2013 Nov 27. PMID 24288340
- [Background] Tamura M, Shimizu Y, Hashizume Y. Pain following thoracoscopic surgery: retrospective analysis between single-incision and three-port video-assisted thoracoscopic surgery. J Cardiothorac Surg. 2013 Jun 12;8:153. doi: 10.1186/1749-8090-8-153. PMID 23759173
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Tulgar S, Senturk O. Ultrasound guided low thoracic erector spinae plane block for postoperative analgesia in radical retropubic prostatectomy, a new indication. J Clin Anesth. 2018 Jun;47:4. doi: 10.1016/j.jclinane.2018.02.013. Epub 2018 Mar 5. No abstract available. PMID 29518667
- [Background] Wang HJ, Liu Y, Ge WW, Bian LD, Pu LF, Jiang Y, Zhu GF, Jin XW, Li J. [Comparison of ultrasound-guided serratus anterior plane block and erector spinae plane blockperioperatively in radical mastectomy]. Zhonghua Yi Xue Za Zhi. 2019 Jun 18;99(23):1809-1813. doi: 10.3760/cma.j.issn.0376-2491.2019.23.012. Chinese. PMID 31207693
- [Background] Wang L, Wang Y, Zhang X, Zhu X, Wang G. Serratus anterior plane block or thoracic paravertebral block for postoperative pain treatment after uniportal video-assisted thoracoscopic surgery: a retrospective propensity-matched study. J Pain Res. 2019 Jul 23;12:2231-2238. doi: 10.2147/JPR.S209012. eCollection 2019. PMID 31413621
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- See also: Clincalc.com opioid equivalent calculator — https://clincalc.com/Opioids/